CLINICAL TRIAL: NCT02159300
Title: Brain Rhythms in Fibromyalgia: A Magnetoencephalography (MEG) Study
Acronym: FMP
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: WS697348
Record Dates: First submitted 2014-06-02; First posted 2014-06-09 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with fibromyalgia pain Intervention: experience brain activity recording
  Interventions: Behavioral: experience brain activity recording
- Healthy Controls: Healthy controls without chronic pain of any type.
  Interventions: Behavioral: experience brain activity recording

INTERVENTIONS:
Behavioral: experience brain activity recording — Intervention: experience brain activity recording
  Other Names: Change in pain level

SUMMARY:
The long-term purpose of the investigator's research is to understand the pathophysiological basis of chronic pain. This will help provide a framework for the development of effective treatments. The purpose of this specific study is to find if there are abnormal brain rhythms in patients with fibromyalgia syndrome (FM) who are in pain since this will indicate particular types of treatments.

FM is a disorder of the muscles and/or joints, and patients experience sever fatigue. FM occurs more often in women than in men (3.4% of women, 0.5% of men). The diseases can appear at any age, but in most of the cases it occurs in women of childbearing age. FM is considered a chronic pain condition since the pain is persistent. Pain and tenderness can be widespread throughout the body. FM patients are more sensitive to sound and pressure stimulation than healthy controls, indicating that there may be changes in the brain. Also, pain is made worse under conditions of stress.

Treatments for FM pain include life style changes such as exercise, dietary changes, cognitive-behavioral therapy, medications and even surgery, but there is no accepted "best" treatment. This is partly because the underlying cause of the pain is not well understood. The design of this study is to record brain activity to find if there are abnormal brain rhythms in people with FM that are not present in healthy adults of the same age.

Specifically, the investigators will test the hypothesis that constant low frequency oscillations will be present in patients with chronic pain due to FM. This has been found in people with other types of pain and is called Thalamocortical Dysrhythmia (TCD). The study has two parts. In the first part, a complete medical history will be obtained, including a description of the person's pain. In the second part the investigators will use magnetoencephalography (MEG) to non-invasively record brain activity. The MEG data will be analyzed in terms the presence of normal alpha rhythm and abnormal low and high frequency oscillations. Each person will have an MRI so the investigators can localize the rhythms recorded by the MEG in the person's brain using their MRI. The people who record and analyze the MEG recordings will not know if the person is a healthy control or a FM patient. The two parts will be joined to test the hypothesis and find if there is a correlation between the people with abnormal low frequency brain rhythms and the presence or degree of pain.

DETAILED DESCRIPTION:
The investigators will use magnetoencephalography (MEG) to non-invasively record brain activity in women with fibromyalgia (FM) pain and in healthy subjects. The MEG data will be analyzed in terms of the presence of normal alpha rhythm and abnormal low frequency and gamma oscillations and their source in the person's brain using their MRI. The investigators will use clinical evaluation, MEG recordings and MRI scans to achieve the following aims:

1. Determine if abnormal brain rhythms in the delta (<4Hz) and theta (4-8Hz) frequency bands are present in patients with FM while they are in pain. The hypothesis predicts that such low frequency activity will be present in FM patients in pain, but not in healthy controls or patients not in pain.
2. To determine if brain activity in the gamma (35-55Hz) frequency range is present in FM patients. The hypothesis predicts that, in FM patients, areas of low frequency activity will have an "edge" area of high frequency activity.
3. To determine if brain activity in the alpha (8-12Hz) frequency range is present in FM patients and it if decreases in MEG recording made with the eyes open compared to recordings with the eyes closed. Such normal activity is expected in both FM patients and healthy controls.
4. To determine the location of the sources generating abnormal brain rhythms and normal alpha rhythms in FM patients in pain and in healthy controls and patients not in pain. The hypothesis predicts that low frequency regions with high frequency 'edges' will have two locations: a) if the pain is localized, the somatosensory cortex in the region of pain, b) the orbitofrontal cortex in portion of the pain pathway associated with the emotional aspects of pain. The source of normal alpha rhythms in both patients and controls will be localized to the posterior brain, particularly the visual cortex.

A multi-disciplinary treatment approach is taken for FM patients. This includes life style changes such as exercise, dietary changes, cognitive-behavioral therapy as well as medications and even surgery. There is no accepted "best" treatment, and not even a "best" medication. This is partly because the underlying cause of the pain is not well understood. The design of this study is to record brain activity to find if there are abnormal brain rhythms in patients with FM that are not present in healthy adults of the same age. Such a finding would inform more direct treatments that would be directed to the cause of the pain, rather then the symptoms.

Recently, abnormal brain connectivity has been reported in FM patients (Napadow et al., 2010). Also, activation of the frontal cortex, motor and cingulate brain regions has been seen in FM patients during pain anticipation that were correlated with the subsequent pain reported (Burgmer et al., 2010).

These results will be considered in the context of a comprehensive clinical evaluation to determine if thalamocortical dysrhythmia (TCD) is present in patients in pain (Jeanmonod, 1993; Llinas et al, 1999, 2001, 2005). The investigators will also find if abnormal brain rhythms are correlated with the presence and degree of pain and if there is a difference between patients in pain and healthy adults.

II. Study Design. The investigators will follow a recent protocol used in our study of abnormal rhythms in complex regional pain syndrome (Walton et al., 2010). Those who meet criteria for inclusion but not exclusion will be enrolled in the study.

III. METHODS AND PROCEDURES

1. Clinical Examination of Patients

   Information collected during the clinical assessment will include:
   * Demographics: age, sex, employment status.
   * A detailed history of fibromyalgia.
   * A review of pain characteristics: location and severity, quality of pain, timing, duration and context of pain, associated signs and symptoms, exacerbating factors, alleviating factors, motor/sensory loss, and effect of activities of daily living.
   * A complete medical history and important family medical history.
   * A social history: tobacco, alcohol, and illicit drug use.
   * A review of all concomitant medications.
   * Vital signs: blood pressure, heart rate, respiratory rate, height, weight.
   * A physical exam.
   * Confirmation of the presence of the American College of Rheumatism's 1990 criteria for fibromyalgia.
   * Completion of the following clinical assessments by the patient:
   * Visual Analogue Scale-average weekly recall of pain
   * Pain Drawing for localization
   * Fibromyalgia Impact Questionnaire
   * Patient's Global Assessment of Fibromyalgia
   * Medical Outcomes Study Sleep Scale
   * Hospital Anxiety and Depression Scale

   Healthy Controls will have the same procedures as the patients; Clinical Screening, MEG and MRI.
2. MEG recordings Informed consent will be obtained before the MEG recording. If it has been obtained, this will be confirmed. (A member of the study team will bring a copy of the signed informed consent before the MEG recording session.)

   The head shape, including the location of the three fiducial markers (left and right preauricular points, and the nasion) will be obtained for each subject using a 3D tracking system by moving a stylus to each fiducial point and over the surface of the head (Fastrak, Polhemus, Colchester, VT).

   Each participant will be seated in the MEG instrument that is located inside a multi-layer mu-metal magnetically shielded room. The location of the head will be monitored at the beginning and end of each run using electrodes attached to the three fiducial marker points used to obtain the head shape. Head position changes up to ≈0.5 cm will be accepted. (The same fiducial points will be used for the MRI to co-register the MEG and MRI data.)

   Each person will have three MEG recording sessions. Two MEGs will be recorded with the eyes closed (EC), and one will be recorded with the eyes open (EO). Including the time to fill out paperwork, measure their head shape, and the time between MEG recordings, the investigators estimate that each participant will spend 60-90 minutes at the New York University Center for Neuromagnetism.

   Instructions to participants for MEG recordings. An investigator will explain that the purpose of the recording is to look at brain activity while the patient is relaxed. There will be three 7-minute recordings. The first will be with the eyes closed. They will be told to please relax, but try not to fall asleep. Next, there will be a recording period with the eyes open. They will be told to please try not to move the eyes, but look at something the entire time. Third, there will another recording with the eyes closed. The investigator will let the person know when the recording begins, half way through each recording, and come in to see how they are doing after each recording. The person will be asked to please try not to move the head during the recordings.

   Magnetoencephalography is FDA approved and is routinely used for brain mapping in epilepsy and in pre-surgical patients and is standard of care in these cases (Shiraishi et al., 2005; Makela et al., 2006). However, these recordings are being performed exclusively for research purposes. Magnetic fields will be recorded using a 275-channel whole-head MEG system (CTF Systems Inc., Port Coquitlam, British Columbia, Canada) (McCubbin et al., 2004). A third-order software gradient (Weinberg et al., 1984) will be used with a recording bandpass of 0.25-125 Hz.
3. Data Analysis and Data Monitoring. During each run magnetic fields will be recorded in 42 consecutive 10-sec trials. In this way, if the person moves during the session, the 10 sec trial during which this occurs can be eliminated from analysis. Neuromagnetic fields will be recorded in the eyes-closed state to minimize signals from ocular muscles and high-frequency visual system activation, and in the eyes-open and fixated state to decrease the amplitude of the alpha-range (8-12 Hz) peak (and thereby better facilitate the examination of spectrally proximal signals). Spectral analysis and independent component analysis will be carried out as in our previous studies (Walton et al, 2010).

MRI and Source Reconstruction The purpose of the MRI (without contrast) is to provide an anatomical image of the person's brain that will be used to localize the brain activity recorded by the MEG. The MEG and MRI recordings must be co-registered so that they can be aligned accurately. The same location markers, called fiducial markers (see above), must be used for the MEG and the MRI. So, it is best if both recordings are done on the same day. The MRI is after the MEG because the MEG instrument can detect magnetic field as small as 10-15 Tesla. The MRI generates a magnetic field that, although small, can be detected by the MEG instrument and interferes with recording brain activity. The location of the three MEG fiducials is marked using a fine point magic marker. The person is then escorted to the MRI suit and the 3 MRI fiducials are put on the person using the magic marker points as guides.

All MRI scans will be carried out on the 3 T Alegra platform, due to its better single-to-noise ration (SNR), spatial and spectral resolution, compared with the 1.5 T instruments. Where MRI data is present the investigators will maintain a degree of uniformity across experiments by performing MRI constrained modified minimum norm inverse modeling on each data set. The MRI constrained inverse will be computed by assuming that the current source density is confined to grey matter as segmented from the MRI data. Each subject's MRI is segmented, and a tessellated cortical surface is reconstructed for each hemisphere using the software FreeSurfer (Dale et al., 1999). These cortical surfaces are then sub-sampled to create a sources pace of ~40,000 vertices. The lead field matrix, L, is computed for the dipole moments normal to the cortical surface or for all components.

Potential biases or problems. A potential bias is during analysis of the MEG data. This will be mitigated since the person analyzing the data will be blinded to the pain status of the subject. Study subjects are identified by a code only in all data.

Procedures, situations, or materials that may be hazardous. None.

3. Data Storage and Confidentiality. Trained staff will conduct interviews in a respectful and sensitive manner. Records will be coded, stored and reviewed by participant number only. These coded records will be kept in locked files in locked offices. Access to computer-based data will be restricted by protection codes and login passwords, and all computers will be kept in rooms with restricted access.

ELIGIBILITY:
Inclusion Criteria:

* female from any racial/ethnic background
* general good health, with no serious or unstable medical conditions
* normal or corrected-to-normal vision and hearing
* meets the American College of Rheumatology criteria for the diagnosis of fibromyalgia for at least 1 year
* has had continued presence of pain for more than 50% of the last month
* a score of >1 on the unidimensional 100-cm visual analog scale (VAS) for pain level
* has been on a stable medication regimen for at least 3 weeks, with no change greater than +/- 20% variation on total daily dosage
* 18-70 years of age
* is right handed
* willing to complete all study procedures
* is capable of giving written informed consent

Exclusion Criteria:

* in-patient
* a history of brain abnormalities such as stroke, ventriculomegaly or periventricular white matter abnormalities
* has not been on a stable medication regimen for at least 3 weeks, with any change greater than +/- 20% variation on medication total daily dosage
* has a history of substance abuse
* has the presence of concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc. that causes pain
* has concurrent participation in other therapeutic trials
* pregnant and nursing mothers
* has severe psychiatric illnesses (current schizophrenia, major depression with suicidal ideation, substance abuse within two years)
* or has current major depression. [Depression in these patients will be assessed with the Hospital Anxiety and Depression Scale (HADS). Categorization of fibromyalgia patients with high depressive symptoms is defined as >8 for the HADS
* has contraindications for MRI scanning or MEG recording, including any of the following: cardiac pacemaker, intracranial clips, metal implants, or external clips within 10 mm of the head, metal in eyes, claustrophobia, obesity and/or any other reason leading to difficulty getting in the MEG chair or laying supine in the MRI magnet for up to one hour
* Existence of any other chronic pain conditions, in addition to fibromyalgia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with fibromyalgia pain in the greater New York City area.
  Pain-free women in the greater New York City area.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Spectral Power of brain magnetic activity | Expected average of one week after MEG recoring
  The power of brain activity in the delta, theta, alpha, beta and gamma frequency ranges.

SECONDARY OUTCOMES:
Brain location of electromagnetic sources of activity | Expected average of one month after MRI
  The part of the brain with activity in the delta, theta, alpha, beta, and gamma frequency ranges.

OTHER OUTCOMES:
Pain scores on the Visual Analogue Scale | At time of magnetic recording
  Level of pain during recording using visual analogue scale (1-10) as reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo R Llinas, MD, PhD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Center for the Study & Treatment of Pain, New York, New York
  - NYU School of Medicine; Center for Neuromagnetism, New York, New York

REFERENCES:
- [Background] Burgmer M, Pogatzki-Zahn E, Gaubitz M, Stuber C, Wessoleck E, Heuft G, Pfleiderer B. Fibromyalgia unique temporal brain activation during experimental pain: a controlled fMRI Study. J Neural Transm (Vienna). 2010 Jan;117(1):123-31. doi: 10.1007/s00702-009-0339-1. Epub 2009 Nov 25. PMID 19937376
- [Background] Dale AM, Fischl B, Sereno MI. Cortical surface-based analysis. I. Segmentation and surface reconstruction. Neuroimage. 1999 Feb;9(2):179-94. doi: 10.1006/nimg.1998.0395. PMID 9931268
- [Background] Jeanmonod D, Magnin M, Morel A. Thalamus and neurogenic pain: physiological, anatomical and clinical data. Neuroreport. 1993 May;4(5):475-8. doi: 10.1097/00001756-199305000-00003. PMID 8513122
- [Background] Llinas RR, Ribary U, Jeanmonod D, Kronberg E, Mitra PP. Thalamocortical dysrhythmia: A neurological and neuropsychiatric syndrome characterized by magnetoencephalography. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):15222-7. doi: 10.1073/pnas.96.26.15222. PMID 10611366
- [Background] Makela JP, Forss N, Jaaskelainen J, Kirveskari E, Korvenoja A, Paetau R. Magnetoencephalography in neurosurgery. Neurosurgery. 2007 Jul;61(1 Suppl):147-64; discussion 164-5. doi: 10.1227/01.neu.0000279212.23010.82. PMID 18813173
- [Background] McCubbin J, Vrba J, Spear P, McKenzie D, Willis R, Loewen R, Robinson SE, Fife AA. Advanced electronics for the CTF MEG system. Neurol Clin Neurophysiol. 2004 Nov 30;2004:69. PMID 16012695
- [Background] Napadow V, LaCount L, Park K, As-Sanie S, Clauw DJ, Harris RE. Intrinsic brain connectivity in fibromyalgia is associated with chronic pain intensity. Arthritis Rheum. 2010 Aug;62(8):2545-55. doi: 10.1002/art.27497. PMID 20506181
- [Background] Shiraishi H, Ahlfors SP, Stufflebeam SM, Takano K, Okajima M, Knake S, Hatanaka K, Kohsaka S, Saitoh S, Dale AM, Halgren E. Application of magnetoencephalography in epilepsy patients with widespread spike or slow-wave activity. Epilepsia. 2005 Aug;46(8):1264-72. doi: 10.1111/j.1528-1167.2005.65504.x. PMID 16060938
- [Background] Walton KD, Dubois M, Llinas RR. Abnormal thalamocortical activity in patients with Complex Regional Pain Syndrome (CRPS) type I. Pain. 2010 Jul;150(1):41-51. doi: 10.1016/j.pain.2010.02.023. Epub 2010 Mar 24. PMID 20338687
- [Background] Weinberg H, Brickett PA, Vrba J, Fife AA, Burbank MB. The use of a squid third order spatial gradiometer to measure magnetic fields of the brain. Ann N Y Acad Sci. 1984;425:743-52. doi: 10.1111/j.1749-6632.1984.tb23597.x. PMID 6331246